CLINICAL TRIAL: NCT04347408
Title: Seroprevalence of SARS-Cov-2 Antibodies in Children - a Prospective Multicentre Cohort Study
Brief Title: Seroprevalence of SARS-Cov-2 Antibodies in Children
Status: Completed | Type: Observational
Sponsor: Queen's University, Belfast (Other)
Collaborators: Belfast Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, Thomas Waterfield, Chief Investigator and Academic Clinical Lecturer, Queen's University, Belfast
Other Study IDs: 282617
Record Dates: First submitted 2020-04-07; First posted 2020-04-15 (Actual); Results first posted 2021-08-18 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: COVID; Corona Virus Infection; Multisystem Inflammatory Syndrome in Children
Keywords: antibodies
MeSH Terms: conditions — Coronavirus Infections; pediatric multisystem inflammatory disease, COVID-19 related | interventions — COVID-19 Serological Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Children: Healthy children of healthcare workers between 2 and 15 years of age
  Interventions: Diagnostic Test: Covid-19 Antibody testing (IgG and IgM); Other: Blood Storage
- Paediatric Multisystem Inflammatory Syndrome: Children admitted to hospital with Paediatric Multisystem Inflammatory Syndrome
  Interventions: Diagnostic Test: Covid-19 Antibody testing (IgG and IgM); Other: Blood Storage
- Serious Infection: Children admitted to hospital with serious infections
  Interventions: Diagnostic Test: Covid-19 Antibody testing (IgG and IgM); Other: Blood Storage

INTERVENTIONS:
Diagnostic Test: Covid-19 Antibody testing (IgG and IgM) — Antibody testing for previous exposure to Covid-19
Other: Blood Storage — Storage of blood for multi-omics analysis

SUMMARY:
It is unknown what proportion of healthy children have been exposed to SARS-Cov-2 and how many have antibodies. The aim of this study is to follow a cohort of healthy children over six months and measure their antibodies to SARS-CoV-2.

DETAILED DESCRIPTION:
Coronaviruses are non-segmented positive-stranded RNA viruses with a roughly 30 kb genome. The majority of coronaviruses cause disease in a specific host species but some have infected humans by cross-species transmission. This process has led to a number of severe outbreaks of human disease including severe acute respiratory syndrome (SARS) in 2003 and Middle East respiratory syndrome (MERS) in 2012.

From December 2019 a novel infection "severe acute respiratory syndrome coronavirus 2" (SARS-CoV-2) was identified in the Wuhan region of China. The infection was identified as the causal factor in a growing number of severe cases of pneumonia. This disease was subsequently named coronavirus disease 2019 (COVID-19) by World Health Organisation (WHO). SARS-CoV-2 has been shown to cause severe disease similar to the previous SARS coronavirus from 2003. Severe disease is associated with pneumonia and damage to vital organs including lung, heart, liver, and kidney.

Fortunately SARS-CoV-2 appears to cause only mild, or no, symptoms in children.

The social distancing measures in the United Kingdom include the closure of schools and the cancelling of routine paediatric clinics. These drastic, but necessary, steps are likely to have a profound effect on the well-being of children.

This study is required to determine what proportion of children have been exposed to SARS-Cov-2 and how many, if any, have neutralizing antibodies. The findings from this study could be used to inform public health decisions regarding the re-opening of schools and other services vital to the well-being of children.

In addition the study will recruit children with paediatric multi-system inflammatory syndrome admitted to the Royal Belfast Hospital for Sick Children along with matched controls with other infections.

ELIGIBILITY:
Healthy children of healthcare professionals.

Exclusion Criteria:

Not currently receiving antibiotics, not admitted to hospital within the last seven days, not receiving immunosuppressive drugs and never diagnosed with a malignancy.

Admitted children with paediatric multisystem inflammatory syndrome and admitted children with other serious infections.

Ages: 1 Month to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged from 0 to 15 who are resident in the United Kingdom
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2023-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Waterfield, BMBCh, Principal Investigator — Queen's University, Belfast
Locations (5):
- United Kingdom (5):
  - Royal Belfast Hospital for Sick Children, Belfast
  - University Hospital of Wales, Cardiff
  - Royal Hospital for Children, Glasgow
  - Public Health England, London
  - Public Health England, Manchester

REFERENCES:
- [Derived] Waterfield T, Watson C, Moore R, Ferris K, Tonry C, Watt A, McGinn C, Foster S, Evans J, Lyttle MD, Ahmad S, Ladhani S, Corr M, McFetridge L, Mitchell H, Brown K, Amirthalingam G, Maney JA, Christie S. Seroprevalence of SARS-CoV-2 antibodies in children: a prospective multicentre cohort study. Arch Dis Child. 2021 Jul;106(7):680-686. doi: 10.1136/archdischild-2020-320558. Epub 2020 Nov 10. PMID 33172887

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 1042 potential participants were screened for inclusion, of whom 50 were excluded; 18 were outside the specified age range, 1 met specific exclusion criteria,16 declined consent and 15 did not undergo phlebotomy. In total 992 were enrolled.
Period: Overall Study
Arm/Group | Healthy Children
Started | 992
Completed | 992
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Children
Number analyzed (Participants) | 992
Age, Continuous [Median (Full Range); unit: years] | 10.1 [2.03 to 15.99]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 483
  Male | 509
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Immunoglobulins (G and M) to SARS-Cov2 in Plasma
Description: • Mean antibody titres (IgG/Total antibody) to SARS-CoV-2 in plasma using ROCH/ABBOTT and DIASORIN assays
Time Frame: 6 months
Population: Healthy children of healthcare workers between 2 and 15 years of age
Measure: Mean (95% Confidence Interval); unit: Titres
Arm/Group | Healthy Children
Number analyzed (Participants) | 992
Titres
  Abbott SARS-CoV-2 IgG Assay (Index S/C) | 4.86 [4.28 to 5.45]
  Elecys Roche SARS-CoV-2 (Cut-Off-Index COI) | 65.32 [43.24 to 87.40]
  Diasorin Liason SARS-CoV-2 IgM (arbitrary units A/U) | 64.17 [37.99 to 90.36]

2. Secondary Outcome: Echocardiogram Ejection Fraction
Description: Measure of cardiac function
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2023-12

3. Secondary Outcome: High-sensitivity Cardiac Troponin Test
Description: Cardiac Enzyme
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2023-12

4. Secondary Outcome: Brain Natriuretic Peptide
Description: Cardiac enzyme
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2023-12

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious and other adverse events were not monitored/assessed.
Description: All-cause mortality, serious and other adverse events were not monitored/assessed.
Groups:
- All-cause Mortality, Serious and Other Adverse Events Were Not Monitored/Assessed.: All-cause mortality, serious and other adverse events were not monitored/assessed.
Arm/Group | All-cause Mortality, Serious and Other Adverse Events Were Not Monitored/Assessed.
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The limitations of this study are that all of the children in this study had only mild disease making comparison between severe and mild disease impossible. The children were also recruited from healthcare workers and the prevalence of antibodies is likely to be lower in the general population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT04347408/Prot_SAP_001.pdf